CLINICAL TRIAL: NCT02428335
Title: Evaluation of Technetium-99m Sestamibi to Determine Muscle Energy Metabolism in RCC (Renal Cell Cancer) Patients Treated With Sunitinib
Brief Title: Study of Muscle Energy Metabolism in RCC Patients Treated With Sunitinib
Status: Withdrawn | Type: Observational
Why Stopped: Insufficient financial resources to conduct research and complete trial.
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Sestamibi 1.0
Record Dates: First submitted 2015-04-21; First posted 2015-04-28 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Renal Cell Cancer; Fatigue
MeSH Terms: conditions — Carcinoma, Renal Cell; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Sunitinib is a chemotherapy approved by the FDA as a standard of care treatment for renal cell carcinoma (RCC). Fatigue is a very common side effect of sunitinib that frequently causes dose reductions. The cause of this fatigue remains unclear. This study will use a special type of scan to study sunitinib-induced fatigue in relation to exercise.

DETAILED DESCRIPTION:
Sunitinib, a type of tyrosine kinase inhibitor (TKI) has been approved by the FDA as a standard of care treatment for renal cell carcinoma (RCC). Fatigue is a very common side effect of sunitinib that frequently causes dose reductions. The cause of this fatigue remains unclear. It has been shown that TKIs disrupt growth factor pathways in muscles leading to muscle shrinkage. If sunitinib associated fatigue is due to altered muscle physiology at a molecular level, there will be observable changes in the uptake of 99mTc-sestamibi in scintigraphy scans. The study objective is to determine if sunitinib-induced fatigue as determined by VO2 and QOL fatigue related questionnaire responses are correlated to molecular changes in the muscles as evidenced by 99mTc-sestamibi uptake.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent before any study procedures completed
2. Patients must have histologically or cytologically confirmed RCC.
3. Four weeks must have elapsed since prior chemotherapy, hormonal therapy, targeted therapy or radiation therapy. There is no restriction on the amount of bone marrow previously radiated.
4. Recovery to baseline or, at most, grade 1 of all drug-related toxicities due to prior chemotherapy, radiation, hormonal therapy, or molecular targeted therapy, expect for alopecia.
5. Male / female subject ≥ 18 years of age
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of <2 (Karnofsky >70%)
7. Life expectancy of at least 12 weeks
8. Normal organ and marrow function as defined by :

   * absolute neutrophil count (ANC) > 1500/mcL
   * hemoglobin (Hb) > 90 g/L
   * platelet count ≥ 1000.000/mcL,
   * total bilirubin ≤ 1.5 x the upper limit of normal range (ULN)
   * alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x ULN (<5 x ULN presence of liver metastases)
   * creatinine < 1.5 x institutional ULN
9. Cardiac ejection fraction by MUGA scan or echocardiogram must be >50% for patients at baseline.
10. Ability to understand the purpose of the study and the willingness to sign a written informed consent document
11. Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment. Standard Nuclear Medicine department pregnancy screening will be conducted prior to each 99mTc-sestamibi scan. Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation. The investigator is requested to advise the patient how to achieve an adequate contraception.
12. Patients must give written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.

Exclusion Criteria:

1. Patients who have had chemotherapy, hormonal therapy, molecular targeted therapy, or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
2. Patients may not be receiving any other investigational agents, chemotherapy, immunotherapy, radiotherapy, or molecular targeted agents.
3. Prior treatment with a drug with known anti-angiogenic properties, including other tyrosine kinase inhibitors to VEGFR
4. Any psychological, familial, sociological, or geographical conditions that do not permit medical follow-up and compliance with the study protocol.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, HIV, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Patients that are on therapeutic dose of coumadin or an INR of 1.5 c ULN. Patients that are on low dose coumadin (2mg or less for patency of the central venous catheter) or therapeutic dose of low molecular weight heparin will be allowed.
7. Patients who cannot swallow
8. Patients who are breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women aged 18 years of age or older with a confirmed diagnosis of renal cell carcinoma. Participants will receive standard of care treatment with sunitinib. Participants must be willing to undergo exercise testing and diagnostic imaging with technitium 99m-sestamibi
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
99mTc-sestamibi uptake in muscle cells | 12 weeks from start of treatment
99mTc-sestamibi uptake in muscle cells | 24 weeks from start of treatment
99mTc-sestamibi uptake in muscle cells | 36 weeks from start of treatment

SECONDARY OUTCOMES:
Incidence of sunitinib related fatigue | 36 weeks after the start of sunitinib treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sawyer, MD, Principal Investigator — Alberta Health services
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada